CLINICAL TRIAL: NCT00298246
Title: Clinical and Immunological Investigations of Subtypes of Autism
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060102; 06-M-0102
Record Dates: First submitted 2006-03-01; First posted 2006-03-01 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-03-15

CONDITIONS: Autism Spectrum Disorders; Seizures
Keywords: Neurodevelopmental Disorders; Neurological Disorder; Children- Onset; Children; Pervasive Developmental Disorder; PDD; Autism; Healthy Volunteer; HV
MeSH Terms: conditions — Autism Spectrum Disorder; Seizures; Neurodevelopmental Disorders; Nervous System Diseases; Child Development Disorders, Pervasive; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to learn more about autism and its subtypes. Autism is a developmental disorder in which children have problems with communication and social skills and display restricted interests and repetitive behaviors.

This study has several goals. One aim is to look at types of autism that are known, such as the regressive subtype, (where skills are lost). We will explore whether there is a unique change in immune functioning related to this subtype. Another aim is to serve as one of the sites that will pilot a larger natural history study, entitled Autism Phenome Project. The goal is to further understand autism by identifying other subtypes.

We will look at several types of medical issues that may be related to autism, including immunologic problems. Children will be followed over the course of several years. We aim to capture medical problems that may be related to autism as they develop, and study outcomes in areas such as behavior and language, in order to explore known and new subtypes of autism.

Normally developing children (aged 1) with autism (age 1, and developmental delays other than autism (age 1), may be eligible for this study.

Depending on each child's study group and age, participants may undergo the following tests and procedures:

Baseline Visit

* Medical and developmental history, physical examination, psychological, cognitive and medical tests to assess symptoms of autism or other developmental disorders, photographs of the child's face, collection of hair, urine and baby teeth samples. If available, hair samples from the baby's first haircut and from the biological mother's hair are also collected.
* Overnight electroencephalogram (EEG): A special cap with electrodes is placed on the child's head to measure brain waves (brain electrical activity) while the child sleeps in the hospital overnight. Healthy volunteers do not undergo this procedure.
* Magnetic resonance imaging (MRI) scan: The child stays in the scanner, lying still for 10 to 15 minutes at a time. Since it may be difficult for the child to lie still, the test may be scheduled for a time when the child is likely to be sleepy, or the child may be sedated.
* Lumbar puncture (for children in the autism). This test and the MRI may be done under sedation.

Follow-Up Visits

Follow-up visits are scheduled at different intervals, depending on study group, age and aspect of the study the child is enrolled in. The visits include a short interview session with the child's caregiver and assessment of the child's development and behavior. Some of the assessment measures used during the baseline examination are repeated, including symptoms ratings, behavioral tests and a blood test. For some children, the final visit will include repeats of the medical procedures.

DETAILED DESCRIPTION:
Objective:

The current investigation focuses on finding meaningful subtypes of autism. Our objectives include using comprehensive and longitudinal medical assessments and behavioral testing to find subgroups of children with autism with profiles that comprise distinct biological/behavioral phenotypes.

Specific goals include determining if there is a unique alteration in immune function among autistic children with a regressive clinical course, and identifying autism-specific sleep and electroenchelalogram (EEG) abnormalities, and other potential biomarkers.

Study Population:

We are conducting a longitudinal natural history study of 140 children with autism, 12 to 84 months of age at study entry. We also are following as many as 75 typically developing children, and 50 children with Developmental Delay to serve as age-/sex-matched controls.

Design:

Systematic prospective evaluations are being utilized to determine diagnostic and functional outcomes, and evaluate behavioral, medical and immunologic functioning. These evaluations include comprehensive medical history, behavioral assessment, physical and neurologic examination, polysomnography (PSG) and EEG, and blood work for laboratory assays. Baseline evaluations also included MRI and lumbar puncture (the latter was only subjects with autism). In any investigation of behavioral outcomes and potential biomarkers, repeated assessments are necessary to determine whether findings are due to state versus trait alterations. Thus, key elements of the assessments are repeated every 6 to 12 months, depending on the child s age.

Outcome Variables:

Measures of autism symptoms and severity, along with cognitive and adaptive behavior profiles, will be used as behavioral outcome variables.

Results of physical and neurological examinations, genetic testing, EEGs, polysomnograms, MRI scans and laboratory assays of blood and CSF will be tested for their utility as biomarkers of autism s core symptoms or identification of etiologically related subgroups of patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* There are 3 participant groups in this study.

  * AUT: Children with autism (diagnosed with autistic disorder according to DSM-IV criteria). This group will include children that may be dichotomized as with regression and without regression.
  * DD: Children with nonspectrum developmental delays
  * TYP: Children deemed to be typically developing
  * Accrual numbers are to include 140 children in the AUT group, 50 children in the DD group and 75 children in the TYP group.
* AUT: Children are included if they meet DSM-IV criteria for autistic disorder, based on ADI-R and ADOS and clinical judgment. Those meeting research criteria for autism will be included.
* Regression is defined as: Language loss: Loss of at least 3 spontaneously meaningful words (excluding mama or dada) used for at least a month, and lost for at least a month.AND/OR Nonverbal communication/social loss: Loss of more than one nonverbal communicative behavior (e.g. gestures, joint attention, eye contact, imagination, pretend play, sharing, showing, watching children, orienting to name, social smiling, social games, spontaneous imitation of actions, response to social overtures). Although there is overlap in the age period for regression specified in this protocol (regression between 15-30 months) and that described for childhood disintegrative disorder (CDD) (the DSM-IV criteria for indicate apparently normal development for the first 2 years after birth ), the criteria for CDD also indicate a diagnosis can only be made if symptoms are not better accounted for by another pervasive developmental disorder such as autism. Symptoms of CDD that separate it from autism include loss of acquired skills in areas such as motor skills and bowel or bladder control, while the focus of the current study is on regression in core symptoms of autism (i.e. socio-communicative skills). Thus, the currently protocol will include children with regression over 2 who meet criteria for autism, but not those who only meet criteria for CDD.
* DD: Developmental scores (Performance Quotient and Verbal Quotient) greater than 1.5 standard deviations below mean on Mullen Scales of Early Learning
* TYP: No diagnosis of developmental delay, and no first-degree relatives with a history of autism spectrum disorders.

EXCLUSION CRITERIA:

* Diagnosis of cerebral palsy. For the typical controls only, a history of extremely low birth weight (due to prematurity or intrauterine growth failure).
* If behavioral management issues (e.g. self-injury, aggressiveness) are severe to the extent that the screening protocol was aborted.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 557 (Actual)
Dates: Start 2006-02-22; Study Completion 2017-03-15

PRIMARY OUTCOMES:
Behavioral profiles | 6 to 12 months
Immune markers | 6 to 12 months
Sleep/EEG findings | 6 to 12 months
Neuroimaging findings | 6 to 12 months
Other laboratory findings | 6 to 12 months
Genetic abnormalities | 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahlsen G, Rosengren L, Belfrage M, Palm A, Haglid K, Hamberger A, Gillberg C. Glial fibrillary acidic protein in the cerebrospinal fluid of children with autism and other neuropsychiatric disorders. Biol Psychiatry. 1993 May 15;33(10):734-43. doi: 10.1016/0006-3223(93)90124-v. PMID 8353169
- [Background] Ashwood P, Anthony A, Pellicer AA, Torrente F, Walker-Smith JA, Wakefield AJ. Intestinal lymphocyte populations in children with regressive autism: evidence for extensive mucosal immunopathology. J Clin Immunol. 2003 Nov;23(6):504-17. doi: 10.1023/b:joci.0000010427.05143.bb. PMID 15031638
- [Background] Ashwood P, Van de Water J. Is autism an autoimmune disease? Autoimmun Rev. 2004 Nov;3(7-8):557-62. doi: 10.1016/j.autrev.2004.07.036. PMID 15546805
- [Derived] Farmer CA, Thurm AE, Honnekeri B, Kim P, Swedo SE, Han JC. The contribution of platelets to peripheral BDNF elevation in children with autism spectrum disorder. Sci Rep. 2021 Sep 13;11(1):18158. doi: 10.1038/s41598-021-97367-4. PMID 34518555
- [Derived] Tierney E, Remaley AT, Thurm A, Jager LR, Wassif CA, Kratz LE, Bailey-Wilson JE, Bukelis I, Sarphare G, Jung ES, Brand B, Noah KK, Porter FD. Sterol and lipid analyses identifies hypolipidemia and apolipoprotein disorders in autism associated with adaptive functioning deficits. Transl Psychiatry. 2021 Sep 9;11(1):471. doi: 10.1038/s41398-021-01580-8. PMID 34504056
- [Derived] Oztan O, Garner JP, Partap S, Sherr EH, Hardan AY, Farmer C, Thurm A, Swedo SE, Parker KJ. Cerebrospinal fluid vasopressin and symptom severity in children with autism. Ann Neurol. 2018 Oct;84(4):611-615. doi: 10.1002/ana.25314. Epub 2018 Sep 26. PMID 30152888
- [Derived] Manwaring SS, Mead DL, Swineford L, Thurm A. Modelling gesture use and early language development in autism spectrum disorder. Int J Lang Commun Disord. 2017 Sep;52(5):637-651. doi: 10.1111/1460-6984.12308. Epub 2017 Jan 24. PMID 28120370
- [Derived] Pardo CA, Farmer CA, Thurm A, Shebl FM, Ilieva J, Kalra S, Swedo S. Serum and cerebrospinal fluid immune mediators in children with autistic disorder: a longitudinal study. Mol Autism. 2017 Jan 5;8:1. doi: 10.1186/s13229-016-0115-7. eCollection 2017. PMID 28070266
- [Derived] Shoffner J, Trommer B, Thurm A, Farmer C, Langley WA 3rd, Soskey L, Rodriguez AN, D'Souza P, Spence SJ, Hyland K, Swedo SE. CSF concentrations of 5-methyltetrahydrofolate in a cohort of young children with autism. Neurology. 2016 Jun 14;86(24):2258-63. doi: 10.1212/WNL.0000000000002766. Epub 2016 May 13. PMID 27178705
- [Derived] Thurm A, Himelstein D, D'Souza P, Rennert O, Jiang S, Olatunji D, Longo N, Pasquali M, Swedo S, Salomons GS, Carrillo N. Creatine Transporter Deficiency: Screening of Males with Neurodevelopmental Disorders and Neurocognitive Characterization of a Case. J Dev Behav Pediatr. 2016 May;37(4):322-6. doi: 10.1097/DBP.0000000000000299. PMID 27096572
- [Derived] Smith E, Thurm A, Greenstein D, Farmer C, Swedo S, Giedd J, Raznahan A. Cortical thickness change in autism during early childhood. Hum Brain Mapp. 2016 Jul;37(7):2616-29. doi: 10.1002/hbm.23195. Epub 2016 Apr 7. PMID 27061356
- [Derived] Buckley AW, Scott R, Tyler A, Mahoney JM, Thurm A, Farmer C, Swedo S, Burroughs SA, Holmes GL. State-Dependent Differences in Functional Connectivity in Young Children With Autism Spectrum Disorder. EBioMedicine. 2015 Nov 5;2(12):1905-15. doi: 10.1016/j.ebiom.2015.11.004. eCollection 2015 Dec. PMID 26844269
- [Derived] Lane R, Kessler R, Buckley AW, Rodriguez A, Farmer C, Thurm A, Swedo S, Felt B. Evaluation of Periodic Limb Movements in Sleep and Iron Status in Children With Autism. Pediatr Neurol. 2015 Oct;53(4):343-9. doi: 10.1016/j.pediatrneurol.2015.06.014. Epub 2015 Jun 26. PMID 26231264
- [Derived] Thurm A, Manwaring SS, Swineford L, Farmer C. Longitudinal study of symptom severity and language in minimally verbal children with autism. J Child Psychol Psychiatry. 2015 Jan;56(1):97-104. doi: 10.1111/jcpp.12285. Epub 2014 Jun 24. PMID 24961159
- [Derived] Graf-Myles J, Farmer C, Thurm A, Royster C, Kahn P, Soskey L, Rothschild L, Swedo S. Dietary adequacy of children with autism compared with controls and the impact of restricted diet. J Dev Behav Pediatr. 2013 Sep;34(7):449-59. doi: 10.1097/DBP.0b013e3182a00d17. PMID 24042076
- [Derived] Joseph L, Thurm A, Farmer C, Shumway S. Repetitive behavior and restricted interests in young children with autism: comparisons with controls and stability over 2 years. Autism Res. 2013 Dec;6(6):584-95. doi: 10.1002/aur.1316. Epub 2013 Jul 18. PMID 23868881